CLINICAL TRIAL: NCT00240656
Title: Official Title: Spironolactone Combined With Captopril and Carvedilol for the Treatment of Patients With Pulmonary Arterial Hypertension Associated With Congenital Heart Disease-Focus on Pulmonary Artery Remodeling
Brief Title: Spironolactone Combined With Captopril and Carvedilol for the Treatment of Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0510-A
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2005-10

CONDITIONS: Hypertension, Pulmonary
Keywords: aldosterone antagonists, spironolactone, captopril carvedilol
MeSH Terms: conditions — Hypertension, Pulmonary

INTERVENTIONS:
Drug: spironolactone captopril carvedilol

SUMMARY:
The purpose of this study is to determine whether a larger dose of the aldosterone antagonist spironolactone combined with an ACE inhibitor (captopril) and a beta-blocker (carvedilol) is effective in reverse pulmonary artery remodeling in patients with pulmonary arterial hypertension (PAH)secondary to congenital heart disease

DETAILED DESCRIPTION:
The pathogenesis of PAH involves multiple mechanisms. However, three common factors are thought to cause the increased pulmonary vascular resistance that characterizes this devastating disease: vasoconstriction, pulmonary vascular proliferation and remodeling, and thrombosis in situ. Advances in our knowledge of the molecular mechanisms involved in PAH suggest that endothelial dysfunction with chronic impaired production of vasoactive mediators plays a key role. Reduced production of vasoactive mediators, such as nitric oxide (NO) and prostacyclin, along with prolonged overexpression of vasoconstrictors such as endothelin-1 (ET-1), not only affect vascular tone but also promote vascular remodeling. Thus, these substances represent logical pharmacological targets. Animal studies showed ET-1 could stimulate aldosterone secretion in different species, both in vivo and in vitro. This stimulation involves the ET-B alone and both ET-A and ET-B receptor subtypes in rats and humans. Animal studies also showed spironolactone combined with ACE inhibitor could normalize blood pressure, prevents upregulation of vascular ET-1, restore nitric oxide (NO)-mediated endothelial dysfunction. Beta-blockers have ability to reduce dp/dt in pulmonary artery, as well as left ventricle, thus prevent further damage to the dysfunctional endothelium. Furthermore, we observed from our practice that the aforementioned therapy could lower pulmonary artery pressure in patents with pulmonary hypertension secondary to left ventricular dysfunction. Thus, we hypothesize spironolactone combined with ACE inhibitor and beta-blocker has the ability to reverse remodeling of pulmonary artery in PAH patients.

ELIGIBILITY:
Inclusion Criteria:

* A mean pulmonary artery pressure higher than 25 mm Hg or, when estimated by echocardiography, pulmonary artery pressure more than half the systemic artery pressure
* Congenital systemic-to-pulmonary shunts

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-10; Study Completion 2006-05

PRIMARY OUTCOMES:
Dyspnoea score
Exercise capacity (six-minute walk)
NYHA/WHO functional class
Change of acropachy
Blood gas test
Pulmonary artery pressure (measured by echocardiogram or catheter)

SECONDARY OUTCOMES:
Other echocardiographic changes:
Systolic pulmonary arterial pressure
Change of right to left shunt expressed by time-velocity integral (TVI) from the defect
Change of left to right shunt expressed by TVI from the defect
Right ventricular (RV) acceleration time (ms)
RV ejection time (ms)
Ratio of RV ejection time/RV acceleration time
Pulmonary arterial valve TVI
Change of diameters of both left and right ventricles
Change of diameters of both left and right atrium
Doppler mitral valve (MV) TVI
Blood gas test

CONTACTS AND LOCATIONS:
Overall Officials: Kunshen Liu, M.D., Study Chair — The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China